CLINICAL TRIAL: NCT07284407
Title: Effects of Pain Neuroscience Education With Sensory Discrimination Training on Pain Catastrophizing, Kinesiophobia and Functional Movements Among Patients With Chronic Low Back Pain: A Randomized Controlled Trial
Brief Title: Effects of Pain Neuroscience Education With Sensory Discrimination Training Among Patients With Chronic Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore University of Biological and Applied Sciences (Other)
Responsible Party: Principal Investigator, Dr. Muhammad Tariq Rafiq, Associate professor, Lahore University of Biological and Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UBAS/ERB/FoRS/25/028
Record Dates: First submitted 2025-11-17; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Low Back Pain
Keywords: Pain Catastrophizing; Kinesiophobia; Functional movements; Neuroscience pain education
MeSH Terms: conditions — Low Back Pain; Kinesiophobia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Participants in the experimental group will receive a 45-minute intervention session consisting of three integrated components (Pain Neuroscience Education, Core Stability Exercises and Graded Sensory Discrimination Training )
  Interventions: Other: Pain Neuroscience Education with Sensory Discrimination Training and Core Stability Exercises
- Control group (Active Comparator): Participants in the control group will receive the same 45-minute sessions consisting of two components (Pain Neuroscience Education and Core Stability Exercises).
  Interventions: Other: Pain Neuroscience Education and Core stability Exercises

INTERVENTIONS:
Other: Pain Neuroscience Education with Sensory Discrimination Training and Core Stability Exercises — Although both Pain Neuroscience Education and Sensory Discrimination Training have demonstrated potential benefits individually, there is a paucity of research evaluating their combined effects. Integrating cognitive (PNE) and sensorimotor (SDT) approaches may produce synergistic effects, improving pain modulation, functional capacity, and psychological resilience.
  Arms: Experimental Group
Other: Pain Neuroscience Education and Core stability Exercises — Participants in the control group will receive the same 45-minute sessions twice per week, but will not receive sensory discrimination training.
  Arms: Control group

SUMMARY:
The current study is a double-blind, parallel-group randomized controlled trial involving 80 participants with chronic low back pain. The trial will compare a program of Pain Neuroscience Education plus Sensory Discrimination Training and core stability exercises with a program of Pain Neuroscience Education and core stability exercises alone. Interventions will be delivered twice weekly for eight weeks. The primary outcome is pain catastrophizing. Secondary outcomes include kinesiophobia and functional movements. Assessments will be conducted at baseline, 4, and 8 weeks. The trial will be carried out at Nutricao Lahore Clinic and Model Town Hospital, Lahore. The hypothesis is that Pain Neuroscience Education with Sensory Discrimination Training will result in greater reductions in pain catastrophizing and kinesiophobia, as well as improvements in functional movements.

DETAILED DESCRIPTION:
Chronic low back pain is a complex condition influenced by biological, psychological, and sensory factors. Pain Neuroscience Education has been shown to reduce maladaptive pain beliefs and improve pain processing, while Sensory Discrimination Training targets altered cortical representation that frequently occurs in chronic pain conditions. Combining these approaches may offer a complementary effect by addressing both cognitive and sensory dimensions of pain.

This study will evaluate the added value of Sensory Discrimination Training when delivered alongside Pain Neuroscience Education and core stability exercises, compared with a control intervention combining Pain Neuroscience Education, and core stability exercises. The trial uses a double-blind, parallel-group randomized controlled design with a total of 80 participants diagnosed with chronic low back pain.

Participants will be randomly assigned to one of two intervention groups. The experimental group will receive structured Pain Neuroscience Education sessions, Sensory Discrimination Training using surface-based tactile discrimination tasks, and a standardized core stability exercise program. The comparison group will receive the same Pain Neuroscience Education protocol, and the same core stability exercise program. Both interventions will be provided twice per week for eight weeks, with each session lasting 45 minutes.

The study aims to investigate whether the addition of Sensory Discrimination Training results in greater improvements in pain-related cognitions, fear-related movement avoidance, and functional movement performance. The primary mechanism of interest is the potential effect of Sensory Discrimination Training on improving cortical sensory mapping, which may contribute to reduced pain catastrophising and improved motor function. Outcome measures will be assessedat baseline, 4, and 8 weeks (end of intervention). The current study will be conducted at Nutricao Lahore Clinic and Model Town Hospital Lahore under standardized procedures to ensure intervention fidelity and consistent delivery across sessions.

ELIGIBILITY:
Inclusion Criteria:

* Age: 19 to 44 Both Genders Mechanical low back pain (duration more than 6 months and less than 2 years) >4/10 Numerical Pain Rating Scale (NPRS)

Exclusion Criteria:

* Pregnancy or post-partum Trauma Psychological Pain Radicular Pain Cancer, tumor, malignancy Neurological Deficit Recent Surgery <1year

Ages: 19 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Pain Catastrophizing | From enrollment to the end of treatment at 8 weeks
  Pain catastrophizing refers to a maladaptive cognitive and emotional response to actual or perceived pain. Pain Catastrophizing is measured by the Pain Catastrophizing Scale. The Pain Catastrophizing Scale is a validated questionnaire used to measure the degree of catastrophic thinking in individuals experiencing pain (Sullivan et al. 1995). The scale consists of 13 items, each representing a different catastrophizing response. For each item, participants rate their experience using a 5-point Likert scale, where 0 = Not at all (the thought or feeling never occurred) and 4 = All the time (the thought or feeling occurred persistently). The total score ranges from 0 to 52, with higher scores indicating greater levels of pain catastrophizing.

SECONDARY OUTCOMES:
Kinesiophobia | From enrollment to the end of treatment at 8 weeks
  Kinesiophobia is a debilitating fear of movement and physical activity due to the belief that movement will cause pain or re-injury. Kinesiophobia is measured by the Tampa Scale for Kinesiophobia. Tampa Scale for Kinesiophobia is the most widely used and validated tool to assess the fear of movement or re-injury. It contains 17 items. Each item is scored using a 4-point Likert scale with 1 = strongly disagree and 4 = strongly agree. Total score ranges from 17 to 68, with higher scores indicating greater kinesiophobia.
Functional Movements | From enrollment to the end of treatment at 8 weeks
  Functional movement refers to the basic movements that people need in daily life to perform normal activities safely and efficiently. These movements involve multiple joints and muscle groups working together in a coordinated way. Functional movements will be assessed using 2D motion analysis through the Kinovea software. Participants will perform two standardized tasks: forward bending and sit-to-stand. All movements will be recorded using a fixed camera positioned at a consistent height (e.g., 1.2 m) and distance (e.g., 2.5 m) from the participant. Kinovea will be used to extract trunk flexion angle, lumbar deviation from the midline, pelvic tilt angle and task completion time. Higher movement quality, reduced deviation, and faster task completion will be interpreted as improved functional performance.

CONTACTS AND LOCATIONS:
Overall Officials: MUHAMMAD TARIQ RAFIQ, Principal Investigator — Lahore University of Biological & Applied Sciences

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: It will be available after the completion of the study.
Access Criteria: Through the corresponding author.